CLINICAL TRIAL: NCT06927557
Title: The Applicability of the Cumberland Ankle Instability Tool in Basketball Athletes: Validity and Reliability Study
Brief Title: The Applicability of the Cumberland Ankle Instability Tool in Basketball Athletes.
Acronym: The CAIT
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Sakarya University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Research Assisstant, Hacettepe University
Other Study IDs: SUBU 3; 13.03.2025- 54/20 (Other: Sakarya University of Applied Sciences)
Record Dates: First submitted 2025-03-18; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: ankle instability; validity study; reliability study
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to evaluate the applicability, validity, and reliability of the Cumberland Ankle Instability Tool (CAIT) in basketball athletes. Given that a significant proportion of injuries in basketball occur in the ankle, our study holds importance for instability assessments conducted in this population. If the Cumberland Ankle Instability Tool is found to be applicable in basketball athletes, it may be utilized in future research.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the applicability, validity, and reliability of the Cumberland Ankle Instability Tool (CAIT) in basketball athletes. Since most injuries in basketball occur in the ankle, our study is significant for assessing instability in this population. If the Cumberland Ankle Instability Tool is found to be applicable in basketball athletes, it may be utilized in future research.

Hypotheses:

H₀ (Null Hypothesis): The Cumberland Ankle Instability Tool is not applicable, valid, or reliable in basketball athletes.

H₁ (Alternative Hypothesis): The Cumberland Ankle Instability Tool is applicable, valid, and reliable in basketball athletes.

The demographic information of the athletes, including height, age, weight, and years of sports experience, will be recorded. The Cumberland Ankle Instability Tool (CAIT) will be created using Google Forms and distributed to the athletes online.

To assess the reliability of the questionnaire, it will be administered twice to the athletes within a 3 to 7-day interval. The following reliability parameters will be calculated:

Internal consistency, Test-retest reliability, Standard error of measurement (SEM), Minimal detectable change (MDC). For validity assessment, the relationship between the Cumberland Ankle Instability Tool (CAIT) and the Foot and Ankle Ability Measure (FAAM) as well as the Identification of Functional Ankle Instability (IdFAI) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 45
* History of ankle sprain
* Participation in basketball training at least once per week

Exclusion Criteria:

* Participation in basketball training at least once per week

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Basketball athletes with a history of ankle sprain, at least one year of basketball experience, and who participate in basketball training at least once per week.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool | Baseline and after one week
  The CAIT, a 9-item scale, was developed by Hiller et al., in 2006 to assess ankle instability. It encompasses aspects such as ankle pain, instability during activities of daily living, foot adaptation during physical movements, and the perception of spatial awareness in the foot (Hiller et al., 2006). The questionnaire is designed to capture the feeling of instability across various activities, including running, walking, jumping, and descending stairs. Scores on the scale range from 0 to 30, with higher scores indicating greater ankle stability and 0 representing the worst possible score indicating severe instability.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | Baseline
  The Foot and Ankle Ability Measure (FAAM) is a self-reported questionnaire designed to assess functional limitations in individuals with foot and ankle disorders. It evaluates a patient's ability to perform daily and sports-related activities.
  Structure of FAAM:
  FAAM consists of two subscales:
  Activities of Daily Living (ADL) Subscale - Includes 21 items assessing functional abilities in everyday activities.
  Sports Subscale - Includes 8 items evaluating performance in sports-related movements.
  Each item is scored using a 5-point Likert scale, ranging from 4 (No difficulty) to 0 (Unable to do it).
  Scoring:
  Each subscale score is calculated as a percentage of the total possible score. Higher scores indicate better foot and ankle function, while lower scores suggest greater disability.
The Identification of Functional Ankle Instability (IdFAI) | Baseline
  The Identification of Functional Ankle Instability (IdFAI) is a self-reported questionnaire designed to assess the presence and severity of functional ankle instability (FAI) in individuals with a history of ankle sprains or instability.
  Structure of IdFAI:
  The questionnaire consists of 10 items that evaluate:
  History of ankle sprains Perceived ankle instability Functional limitations during daily and sports activities Each item is scored on a weighted scale, with higher scores indicating a greater degree of functional ankle instability.
  Scoring:
  The total IdFAI score ranges from 0 to 37. Scores ≥ 11 indicate the presence of functional ankle instability. Higher scores suggest greater severity of instability.